CLINICAL TRIAL: NCT04535336
Title: Effects of the Vitality Acupunch Exercise Program on the Muscle Mass, Muscle Strength, and Sleep Quality of Older Adults With Sarcopenia
Brief Title: Vitality Acupunch Exercise Program for Older Adults With Sarcopenia
Acronym: VA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Kuei-Min Chen, Ph.D., RN., Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-F(II)-20190045(2)
Record Dates: First submitted 2020-08-31; First posted 2020-09-01 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Muscle Mass; Muscle Strength; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitality acupunch (VA) (Experimental): The VA program took 40 minutes to complete and included 3 phases: 1) activating qi and blood (5 movements, 10 minutes): warm-up exercises that allowed the body to accumulate heat and promote flexibility of the joints to loosen up the body, 2) punching meridians (14 movements, 20 minutes): both hands were used to exert a vibrating effect according to the rhythms that stimulate the 14 meridians in the entire body to improve aerobic endurance, and 3) relaxing body and mind (5 movements, 10 minutes): muscle relaxing exercises to rest the body and cease the qi. Participants in the experimental group received the VA program led by the instructors, who were trained an certified by the PI, 3 times per week and 40 minutes per session for 6 months.
  Interventions: Other: Vitality acupunch (VA) exercise program
- Control (Active Comparator): Participants in the control group continued with their daily activities as usual.
  Interventions: Other: Control

INTERVENTIONS:
Other: Vitality acupunch (VA) exercise program — The VA had 3 phases and took 40 minutes to complete.
  Arms: Vitality acupunch (VA)
Other: Control — Participants maintained their daily activities.
  Arms: Control

SUMMARY:
This project was aimed to test the effects of a six-month VA program on the muscle mass, muscle strength, and quality of sleep of institutional older adults with sarcopenia.

DETAILED DESCRIPTION:
A cluster-randomized controlled trial was conducted to test the effects of a six-month VA program on the muscle mass, muscle strength, and quality of sleep of institutional older adults with sarcopenia. Using convenience sampling, 12 long-term care facilities with 114 older adults were recruited, and then cluster-randomized by the facility to a VA experimental or a control group. The experimental group received the VA program led by certified instructors 3 times per week and 40 minutes per session for 6 months; the control group continued with their regular daily activities. One pre-test and two post-tests, 3 months apart, were conducted.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 65 years old
* have been living in the facility for at least 3 months
* intact cognitive function with the Short Portable Mental Status Questionnaire score ≥ 8
* hand-grip strength < 28 kg for men and < 18 kg for women
* calf circumference < 34 cm for men and < 33 cm for women

Exclusion Criteria:

* have spinal cord injury
* have severe cardiovascular or pulmonary diseases
* have musculoskeletal diseases

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Muscle mass | 6 months
  measured by the calf circumference
Muscle strength | 6 months
  measured by the Digital Handgrip Dynamometer (TKK-5101)

SECONDARY OUTCOMES:
Sleep quality | 6 months
  Measured by the Pittsburgh Sleep Quality Index (PSQI): score ranges from 0-21; > 5 indicates clinically significant sleep disruptions.

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Min Chen, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tung HT, Chen KM, Chou CP, Belcastro F, Hsu HF, Kuo CF. Acupunch Exercise Improved Muscle Mass, Hand Grip Strength, and Sleep Quality of Institutional Older Adults with Probable Sarcopenia. J Appl Gerontol. 2023 May;42(5):888-897. doi: 10.1177/07334648221141413. Epub 2022 Nov 30. PMID 36448359